CLINICAL TRIAL: NCT04403139
Title: VZV-specific Tissue Resident Memory T-cells After Shingrix Vaccination
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christine Johnston, Associate Professor: School of Medicine, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009255; R01AG064800 (NIH)
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Varicella Zoster Virus Infection
MeSH Terms: conditions — Varicella Zoster Virus Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: 30-40 year of age (Other)
  Interventions: Drug: Shingrix
- Cohort 2: 70 years of age or older (Other)
  Interventions: Drug: Shingrix

INTERVENTIONS:
Drug: Shingrix — All participants will receive the FDA-approved recombinant zoster (RZV) vaccine (Shingrix) given at the approved dose and schedule.

SUMMARY:
To evaluate the effect of intramuscular RZV vaccine on VZV-specific skin TRM and circulating T-cells

DETAILED DESCRIPTION:
This is an interventional study of vaccination related to infection with varicella zoster virus. We will enroll participants of two age groups. Cohort 1 will be persons between the ages of 30-40; Cohort 2 will be persons who are 70 years of age or older. All participants will receive the FDA-approved recombinant zoster (RZV) vaccine (Shingrix) given at the approved dose and schedule.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: 30-40 years of age
* Cohort 2: 70 years of age or older
* HIV seronegative

Exclusion Criteria:

* Previous vaccination with Shingrix (RZV), Zostavax (ZVL, zoster vaccine live), or with the chickenpox vaccine
* VZV seronegative
* Active Hepatitis C infection or active Hepatitis B infection. Persons with serologic evidence of hepatitis C infection that has cleared spontaneously, or with a history of treated hepatitis C with a sustained virologic response, can be enrolled. Persons with a history of resolved hepatitis B infection (negative for hepatitis B surface antigen) can be enrolled
* History of a life-threatening allergic reaction (anaphylactic/anaphylactoid reaction) to any component of the vaccine
* History of receipt of an organ transplant or hematopoietic stem cell transplant
* Significant autoimmune disease such as rheumatoid arthritis, psoriatic arthritis, inflammatory bowel disease, multiple sclerosis, scleroderma, dermatomyositis, or other condition which in the past has required significant immune modifying medication or which has a clinical course that is characterized by relapses
* Has immunosuppression as a result of an underlying illness (e.g. leukemia, lymphoma or other malignant neoplasms) or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy.
* Has long-term use of oral or parenteral steroids (>7 days), or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed)
* Women of child-bearing potential only: pregnant, breastfeeding, or planning to become pregnant 3 months post vaccination
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render biopsies unsafe
* History of coagulopathy or taking medication that may cause bleeding (long term high dose aspirin, heparin, coumadin). Aspirin doses <100 mg daily allowed
* History of keloid formation or excessive scarring
* History of frequent cellulitis or boils (>3 episodes in past 2 years) requiring antibiotic therapy
* Allergy to lidocaine, silver nitrate, or mupirocin
* Has any condition or medical history that would, in the opinion of the site principal investigator place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Level of gE-specific IgG in serum. | up to 1 year after vaccination
  Units will be optical density at 492 nanometers from ELISA.
Level of gE-specific CD4 T cells in blood | up to 1 year after vaccination
  Units will be cells per million CD4+ T cells in blood.
Cytokine profile of gE-specific CD4 T cells in blood | up to 1 year after vaccination
  Units will be percent of gE-reactive T cells expressing single T cell cytokines or combinations of cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Johnston, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington Virology Research Clinic, Seattle, Washington, United States